CLINICAL TRIAL: NCT02154984
Title: A Pilot Study of Time Restricted Diet in Obese/Overweight Pre &Amp; Postmenopausal Women
Brief Title: Time Restricted Diet in Obese or Overweight Pre or Postmenopausal Participants
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study closed due to funding before accrual was met
Sponsor: Northwestern University (Other)
Collaborators: Avon Foundation Center of Excellence (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NU 13CC12; NCI-2014-01094 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STU00091568; NU 13CC12 (Other: Northwestern University); P30CA060553 (NIH)
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Healthy, no Evidence of Disease; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Behavioral (time restricted diet) (Experimental): Participants follow a time restricted diet, which restricts daily eating to an 8 hour time window between 12:00-8:00 pm. Participants are allowed to consume non-caloric beverages (water, black tea, black coffee, diet soda, etc.) during the fasting hours and required to record daily food consumption in the smartphone app for 6 months. Participants are also coached by telephone over approximately 10-15 minutes weekly for 1 month and then biweekly for 5 months.
  Interventions: Behavioral: behavioral dietary intervention; Behavioral: telephone-based intervention; Other: laboratory biomarker analysis

INTERVENTIONS:
Behavioral: behavioral dietary intervention — Follow tRD
Behavioral: telephone-based intervention — Receive coaching calls
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
The purpose of this study is to study the relationships between obesity, hormones and menopausal status, and breast cancer. The researchers would like to study whether a type of nutritional intervention, called a time-restricted diet or tRD, is easy to maintain using a smartphone application; the researchers also want to study the effect that a tRD has on weight control, hormones, and breast tissue. A tRD is a type of diet that requires people to restrict their daily eating to a specific time frame each day. The researchers think that this might be an effective and manageable way to control weight.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Feasibility of fostering adherence to self-monitoring of dietary intake using a smartphone application (app).

II. Feasibility of the goal of following a time-restricted diet.

SECONDARY OBJECTIVES:

I. Identify potential molecular biomarkers and/or signatures to explore its efficacy for the normalization of metabolism.

II. Assess the systemic endocrine effects of a time restricted diet (tRD) intervention in overweight and obese pre and postmenopausal women.

III. Assess weight change following a tRD intervention. IV. Evaluate the effects of a tRD intervention, and identify a specific and reproducible genomic signature, in breast samples obtained by random fine needle aspiration in the tRD study population.

V. Assess the volume of parenchymal enhancement on magnetic resonance imaging (MRI).

OUTLINE:

Participants follow a time restricted diet, which restricts daily eating to an 8 hour time window between 12:00-8:00 pm. Participants are allowed to consume non-caloric beverages (water, black tea, black coffee, diet soda, etc.) during the fasting hours and required to record daily food consumption in the smartphone app for 6 months. Participants are also coached by telephone over approximately 10-15 minutes weekly for 1 month and then biweekly for 5 months.

After completion, participants are followed up for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have a stable weight (have not gained or lost 25 pounds in the last 6 months)
* Subjects must have had a normal mammogram within 9 months prior to registration; NOTE: subjects must also have a normal breast exam on the day of the pre-intervention random fine needle aspiration (rFNA)
* Subjects must have a body mass index (BMI) of 25-40
* Subjects must fit into ONE of the following menopausal categories:

  * Premenopausal (n = 40) - defined as meeting all the following criteria:

    * Have had at least 8 menstrual cycles in the past 12 months
    * Have had no hormonal contraception in the past 3 months prior to registration
    * Have serum hormone parameters (estradiol [E2], progesterone, follicle stimulating hormone [FSH]) in premenopausal range on the day of rFNA; NOTE: subjects will self-report menopausal status at registration, and confirmation of hormonal parameters will occur after registration as part of pre-intervention procedures; if there is mis-assignment of status, the recruitment of future subjects will be adjusted accordingly
  * Postmenopausal (n = 40) - defined as meeting all of the following criteria:

    * Last menstrual period (LMP) > 1 year previously
    * Have had no hormone use in the past 3 months prior to registration
    * Serum E2, progesterone, FSH in postmenopausal range on the day of rFNA; NOTE: subjects will self-report menopausal status at registration, and confirmation of hormonal parameters will occur after registration as part of pre-intervention procedures; if there is mis-assignment of status, the recruitment of future subjects will be adjusted accordingly
* Subjects must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Subjects who have been diagnosed with a prior cancer at any site (other than breast cancer) may participate as long as they have been off medical therapy for at least 12 months prior to registration
* Subjects with prior breast cancer must be off all systemic therapy (including endocrine agents) for at least 2 years prior to registration
* Subjects must be willing to undergo a random fine needle aspiration (rFNA) at the beginning and end of the intervention period
* Subjects must be willing and able to abstain from the use of aspirin for at least 2 weeks prior to undergoing each rFNA procedure (pre- and post-intervention)
* Subjects must have the ability to understand and the willingness to sign a written informed consent prior to registration on study
* Subjects must have a smart phone (newer generation Android or any Iphone) to be able to track their food intake times
* Subjects must be willing to restrict food intake to an 8 hour period every day (12 pm to 8 pm)

Exclusion Criteria:

* Subjects who have received hormonal contraception and/or hormone therapy in the past 3 months are not eligible
* Subjects who are pregnant and/or lactating are not eligible
* Subjects who are noted (upon initial online screening) to do 150 minutes or more of moderate level physical activity each week, get less than 8% of their calories from saturated fat, and eat more than 5 fruit and vegetable servings per day will not be eligible
* Subjects who are part of any structured weight loss programs (e.g. Weight Watchers, etc.) are not eligible
* Subjects who have undergone bariatric surgery are not eligible
* Subjects who work night shifts are not eligible
* Subjects who have diabetes or uncontrolled hypertension are not eligible; NOTE: for the purposes of this study, uncontrolled will be defined as diastolic pressure over 100 mmHg

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-02-23 (Actual); Study Completion 2017-02-23 (Actual)

PRIMARY OUTCOMES:
Adherence to self-monitoring | Up to 3 months after completion of study
  Assessed by demonstrating that at least 65% of participants record dietary intake on at least 80% of study intervention days. Adherence will be assessed via a one-sample chi-squared test for proportions.
Attaining the goal of dietary time restriction | Up to 3 months after completion of study
  Assessed by demonstrating that at least 65% of participants recorded appropriate time restriction on at least 80% of study days.

SECONDARY OUTCOMES:
Changes in steroid hormones (estradiol, progesterone, testosterone) levels | Baseline to up to 3 months after completion of study
  Blood samples will be taken and representative values (mean, standard deviation, median, and range) of hormones and adipokine measurements will be used to calculate changes following intervention, which will then be used for univariate analysis using menopausal status and change in BMI as the main predictors of interest. These analyses are exploratory and descriptive of the systemic endocrine/adipokine environment; they will be related to gene expression changes. Correlations between changes in BMI and changes in biomarker levels will be assessed via the Spearman correlation.
Changes in gonadotropins (FSH) levels | Baseline to up to 3 months after completion of study
  Blood samples will be taken and representative values (mean, standard deviation, median, and range) of hormones and adipokine measurements will be used to calculate changes following intervention, which will then be used for univariate analysis using menopausal status and change in BMI as the main predictors of interest. These analyses are exploratory and descriptive of the systemic endocrine/adipokine environment; they will be related to gene expression changes. Correlations between changes in BMI and changes in biomarker levels will be assessed via the Spearman correlation.
Changes in insulin axis (insulin, insulin-like growth factor 1, IGF binding protein 3, homeostatic model assessment, homocystein) levels | Baseline to up to 3 months after completion of study
  Blood samples will be taken and representative values (mean, standard deviation, median, and range) of hormones and adipokine measurements will be used to calculate changes following intervention, which will then be used for univariate analysis using menopausal status and change in BMI as the main predictors of interest. These analyses are exploratory and descriptive of the systemic endocrine/adipokine environment; they will be related to gene expression changes. Correlations between changes in BMI and changes in biomarker levels will be assessed via the Spearman correlation.
Changes in adipokines (leptin, adiponectin, low molecular weight adiponectin) levels | Baseline to up to 3 months after completion of study
  Blood samples will be taken and representative values (mean, standard deviation, median, and range) of hormones and adipokine measurements will be used to calculate changes following intervention, which will then be used for univariate analysis using menopausal status and change in BMI as the main predictors of interest. These analyses are exploratory and descriptive of the systemic endocrine/adipokine environment; they will be related to gene expression changes. Correlations between changes in BMI and changes in biomarker levels will be assessed via the Spearman correlation.
Changes in inflammatory axis (interleukin-6, tumor necrosis factor alpha) levels | Baseline to up to 3 months after completion of study
  Blood samples will be taken and representative values (mean, standard deviation, median, and range) of hormones and adipokine measurements will be used to calculate changes following intervention, which will then be used for univariate analysis using menopausal status and change in BMI as the main predictors of interest. These analyses are exploratory and descriptive of the systemic endocrine/adipokine environment; they will be related to gene expression changes. Correlations between changes in BMI and changes in biomarker levels will be assessed via the Spearman correlation.
Changes in weight | Baseline to up to 3 months after completion of study
  The pre- and post-intervention measures and within-individual changes in weight be summarized and examined for Normality and outliers; required transformations to achieve Normality will be performed.
Changes in BMI | Baseline to up to 3 months after completion of study
  The pre- and post-intervention measures and within-individual changes in BMI will be summarized and examined for Normality and outliers; required transformations to achieve Normality will be performed. Pre-post comparisons of BMI will be performed using paired Wilcoxon signed-rank tests to evaluate changes over time, designating P < 0.05 as significant.
Changes in breast epithelial gene expression | Baseline to up to 3 months after completion of study
  Gene expression for all 58 genes on the Taqman low density gene expression assays will be summarized to confirm normality and discern outliers. Each gene will then be analyzed using a linear model with the main effect of menopausal status and change in BMI, baseline gene expression and change in expression will be correlated to baseline steroid hormones and adipokines, and their change. If severe departure from normality is observed, these linear models will be applied to ranks of the data.
Changes in parenchymal volume assessed by MRI | Baseline to up to 3 months after completion of study
  The volume of parenchymal enhancement on MRI will be assessed pre and post intervention in women who consent to this optional component.

CONTACTS AND LOCATIONS:
Overall Officials: Seema Khan, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States